CLINICAL TRIAL: NCT05112198
Title: Digital Symptom Tracking, Patient Engagement and Quality of Life in Advanced Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-38423; NCI-2021-12414 (Other: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Quality of Life
Keywords: Patient and clinician engagement; Digital Symptom Tracking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noona web-based symptom tracking tool (Experimental): In addition to usual care for their disease, patients interact with Noona system and system questioners to record their symptoms over a period of 6 months.
  Interventions: Device: Use of Noona web- based symptom tracking tool
- Usual Care (No Intervention): Participants will receive the standard of care for their disease

INTERVENTIONS:
Device: Use of Noona web- based symptom tracking tool — Noona patient reported outcome (PRO) platform tool that summarizes symptoms and distress
  Arms: Noona web-based symptom tracking tool

SUMMARY:
The purpose of this study is to (1) describe patient and clinician engagement in web-based symptom self-monitoring, (2) identify differences in symptom management between intervention and usual care groups, and (3) identify potential outcomes of real-time symptom tracking and management.

With the assistance of the study coordinator, participants randomized to the intervention will create an account with Noona. Patients will be instructed to log symptoms as often as relevant using their own personal devices. Patients will also be prompted once per week for 24 weeks to log any recent symptoms. These participants will be sent a Symptom Questionnaire (SQ) via the Noona tool that summarizes their symptoms and distress one week prior to each oncology clinic visit. Symptoms designated as clinically severe either during regular symptom logging or via the SQ will trigger a prompt to contact the clinical team for immediate follow-up.

DETAILED DESCRIPTION:
New patients from three cancer care programs (thoracic oncology, gastrointestinal oncology, and palliative care) at two academic institutions (Stanford and UCSF) will be screened for demographic and disease stage data within the patient medical record. Eligible patients will be asked by their oncology team whether they would be interested in participating a study of symptom management in oncology care.

Patients who express interest and ability to participate will be interviewed to determine eligibility.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals (men and women) aged 18 years or older
2. Biopsy proven (recurrent or metastatic) advanced lung or gastrointestinal cancer
3. No limit on prior lines of therapy in the metastatic setting
4. ECOG performance status of 0-2
5. Estimated life expectancy of at least 6 months
6. Access to smartphone, tablet or computer with capability to utilize symptom tracking application
7. Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures
8. Willing and able to comply with all study procedures

Exclusion Criteria:

1. Concurrent disease or condition that interferes with participation or safety
2. Non-english speaking, as the application is developed in the english language
3. Non-castrate resistant prostate cancer
4. Enrolled in other non-therapeutic or therapeutic clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with at least one symptom questionnaire (SQ) completed after enrollment using the PROMIS platform | 6 months
Change in PROMIS-G (Patient-Reported Outcomes Measurement Information System-Global) physical subscale score | baseline, 6 months
  Scores goes from (1-5). 5=Excellent and 1=Poor
Change in PROMIS-G (Patient-Reported Outcomes Measurement Information System-Global) mental subscale score | baseline, 6 months
  Scores goes from (1-5). 5=Excellent and 1=Poor

SECONDARY OUTCOMES:
Rate of SQ adherence | 6 months
  Rate of SQ adherence is defined as completing at least 70% of requested SQs
Average number of diary encounters | 6 months
  A Noona system log in is recorded as a diary encounter
Change in overall Functional Assessment of Cancer Therapy-General (FACT-G) score | baseline, 6 months
  Scores goes from (0-4). 4=Very Much and 0=Not at all
Symptom experience | 6 months
  Number of patient-reported symptoms by type and severity
Proportion of clinicians that report satisfactory use of the Noona system | 6 months
Tabulated responses from Noona Patient Feedback questionnaire | 6 months
  Questions include patient response to question about getting started with the Noona system and ease of use and user experience.

CONTACTS AND LOCATIONS:
Overall Officials: Kavitha Ramchandran, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford Cancer Institute, Palo Alto, California
  - UCSF Helen Diller Medical Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: No